CLINICAL TRIAL: NCT06528847
Title: Benmelstobart (TQB2450) for Adjuvant Therapy in Pathologic Stage IB, IASLC Grade 3 Invasive Lung Adenocarcinomas: A Prospective, Single-arm, Phase 2 Clinical Trial
Brief Title: Adjuvant Benmelstobart for Stage IB, Grade 3 Invasive Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Chief Physician, Deputy Head of Thoracic Surgery Dept., Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR010
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Immunotherapy; Adjuvant therapy; Lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Intervention Model Description: This study is a prospective, interventional, single-arm, phase 2 clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Benmelstobart Group (Experimental): Enrolled patients will receive adjuvant immunotherapy with the PD-L1 inhibitor Benmelstobart (TQB2450) at a dose of 1200 mg every 3 weeks by intravenous injection, for a maximum of 16 cycles following radical resection.
  Interventions: Drug: Benmelstobart

INTERVENTIONS:
Drug: Benmelstobart — The PD-L1 inhibitor Benmelstobart (TQB2450) is administered as an adjuvant therapy in patients with pathologic stage IB, IASLC grade 3 invasive lung adenocarcinoma who do not have EGFR active mutations or ALK rearrangement.
  Other Names: TQB2450

SUMMARY:
This study is a prospective, single-arm, phase 2 clinical trial assessing the feasibility, efficacy, and safety of the PD-L1 inhibitor Benmelstobart (TQB2450) as an adjuvant therapy regimen in patients with pathologic stage IB, IASLC grade 3 invasive lung adenocarcinoma without EGFR active mutations or ALK rearrangement.

DETAILED DESCRIPTION:
The target population for this study includes patients with pathologic stage IB, IASLC grade 3 invasive lung adenocarcinoma without EGFR active mutations or ALK rearrangement who have undergone radical resection at Shanghai Pulmonary Hospital. Patients are screened and enrolled within 4 to 12 weeks after surgery. Following surgery, adjuvant chemotherapy may be administered based on the patient's treatment needs or the attending physician's assessment. Subsequently, patients will receive adjuvant immunotherapy with the PD-L1 inhibitor Benmelstobart (TQB2450 injection) at a dose of 1200 mg every 3 weeks by intravenous injection, for a maximum of 16 cycles. The primary endpoint is the 2-year disease-free survival (DFS) rate. The secondary endpoints include the 3-year and 5-year DFS rates, the 5-year overall survival (OS) rate, and drug safety. The sample size is 62 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are able to understand the informed consent form, voluntarily agree to participate, and sign the informed consent form;
2. Participants must be 18 years or older and under 75 years of age on the day they sign the informed consent form;
3. Pathologically confirmed stage IB (AJCC TNM staging, 8th edition) lung adenocarcinoma;
4. Achieved complete resection (R0) after lobectomy, bilobectomy, or sleeve resection;
5. Pathologically diagnosed as grade 3 invasive lung adenocarcinoma according to the 2020 grading system proposed by the International Association for the Study of Lung Cancer (IASLC) Pathology Committee (poorly differentiated: any tumor with 20% or more of high-grade patterns, including solid, micropapillary, and/or complex glandular patterns);
6. No prior receipt of any anti-tumor treatment, including but not limited to systemic chemotherapy, immunotherapy, or radiotherapy;
7. Expected survival time more than 12 weeks;
8. No active EGFR mutations (including but not limited to exon 19 deletions, exon 21 L858R, exon 21 L861Q, exon 18 G719X, or exon 20 S768I mutations) or ALK rearrangements;
9. Tumor PD-L1 expression ≥1% (the PD-L1 IHC 22C3 pharmDx reagent, antibody clone number: 22C3, detection platform: DAKO Autostainer Link 48);
10. Patients are screened and enrolled within 4 to 12 weeks after surgery;
11. Performance status score of 0 or 1 (Eastern Cooperative Oncology Group (ECOG) performance status scale);
12. For female participants of childbearing potential, a negative serum pregnancy test must be obtained within 7 days prior to the first dose of the study drug;
13. Female participants of childbearing potential or male participants with partners of childbearing potential must agree to use highly effective contraception (with an annual failure rate of less than 1%) starting from 7 days before the first dose of the study drug and continuing until 24 weeks after the last dose;
14. Major organ functions must be normal within 7 days prior to the first dose of the study drug.

Exclusion Criteria:

1. Postoperative pathological diagnosis of mixed histological features;
2. Incomplete resection (R1/R2) or wedge resection, segmentectomy;
3. Currently participating in an interventional clinical trial, or having received other investigational drugs or used investigational devices within 4 weeks prior to the first dose of the study drug;
4. Systemic corticosteroids or immunosuppressants must have been administered continuously for 7 days within 14 days prior to the first dose of the study drug;
5. Received live vaccines (including attenuated live vaccines) within 28 days prior to the study drug administration;
6. History of or currently having interstitial lung disease/condition requiring systemic corticosteroid treatment;
7. History of or currently having autoimmune disease;
8. Presence of other malignant tumors within 5 years prior to the first dose of the study drug;
9. Presence of uncontrolled comorbidities such as cardiac, renal, gastrointestinal, or infectious diseases;
10. History of allogeneic bone marrow or organ transplantation;
11. History of using any antibodies or drugs targeting T-cell co-regulatory proteins (immune checkpoints), or previous treatment with anti-tumor vaccines;
12. History of hypersensitivity or intolerance to antibody-based drugs, history of any rapid allergic reactions, uncontrolled asthma, or significant drug allergies;
13. Pregnant and/or breastfeeding women;
14. Other conditions that may affect the safety or compliance of the study drug, including but not limited to psychiatric disorders, uncontrolled large pleural effusions, or moderate to large pleural effusions requiring repeated drainage.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) rate | up to 2 year
  The disease-free survival (DFS) is defined as the time from surgery until disease recurrence, death from any cause, or the end of the study, whichever comes first.

SECONDARY OUTCOMES:
disease-free survival (DFS) rate | up to 3 year
  The disease-free survival (DFS) is defined as the time from surgery until disease recurrence, death from any cause, or the end of the study, whichever comes first.
disease-free survival (DFS) rate | up to 5 year
  The disease-free survival (DFS) is defined as the time from surgery until disease recurrence, death from any cause, or the end of the study, whichever comes first.
overall survival (OS) rate | up to 5 year
  The overall survival (OS) is defined as the time from surgery to death from any cause or the end of the study, whichever comes first.
drug safety | up to 1 year
  The frequency of severe adverse events will be measured from participant enrollment to 30 days after the last drug administration or the initiation of new anti-cancer therapy, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Deping Zhao, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Chang Chen, MD, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng Y, Chen J, Zhang W, Xie C, Hu Q, Zhou N, Huang C, Wei S, Sun H, Li X, Yu Y, Lai J, Yang H, Fang H, Chen H, Zhang P, Gu K, Wang Q, Shi J, Yi T, Xu X, Ye X, Wang D, Xie C, Liu C, Zheng Y, Lin D, Zhuang W, Lu P, Yu G, Li J, Gu Y, Li B, Wu R, Jiang O, Wang Z, Wu G, Lin H, Zhong D, Xu Y, Shu Y, Wu D, Chen X, Wang J, Wang M, Yang R. Benmelstobart, anlotinib and chemotherapy in extensive-stage small-cell lung cancer: a randomized phase 3 trial. Nat Med. 2024 Oct;30(10):2967-2976. doi: 10.1038/s41591-024-03132-1. Epub 2024 Jul 11. PMID 38992123
- [Background] Xue J, Xue L, Tang W, Ge X, Zhao W, Li Q, Peng W, Dai C, Guo Y, Li J. TQB2450 in patients with advanced malignant tumors: results from a phase I dose-escalation and expansion study. Ther Adv Med Oncol. 2024 Jan 6;16:17588359231220516. doi: 10.1177/17588359231220516. eCollection 2024. PMID 38188467
- [Background] Han Y, Wang J, Sun T, Ouyang Q, Li J, Yuan J, Xu B. Predictive biomarkers of response and survival following immunotherapy with a PD-L1 inhibitor benmelstobart (TQB2450) and antiangiogenic therapy with a VEGFR inhibitor anlotinib for pretreated advanced triple negative breast cancer. Signal Transduct Target Ther. 2023 Nov 17;8(1):429. doi: 10.1038/s41392-023-01672-5. PMID 37973901